CLINICAL TRIAL: NCT03200106
Title: Retrospective Study in the Use of the Alfapump and the Treatment of Malignant Ascites
Status: Completed | Type: Observational
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-AAR-011
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Malignant Ascites

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Alfapump — Alfapump implant

SUMMARY:
Treatment of malignant ascites with the alfapump offers a new treatment option for this patient group. So far, there is no systematic analysis of patients with this indication available in the literature.

This retrospective analysis offers the possibility to assemble already existing data within a reasonably short time frame. Based on this analysis, a prospective analysis can be designed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant ascites
* Patients with alfapump implanted for malignant ascites
* Patients 18 years or older at the time of death

Exclusion Criteria:

* Patient is alive at the time of inclusion assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of up to 20 patients' charts who have previously been treated with alfapump will be reviewed.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change in frequency of LVP after implantation of the alfapump | 3-6 months post implant
  The primary objective of the study is to evaluate the performance of the alfapump in reducing the need for large volume paracentesis (LVP) defined as paracentesis of five or more litres of ascites and not by pump paracentesis.

SECONDARY OUTCOMES:
The safety and tolerability of alfapump in patients with malignant ascites | 3-6 months post implant
  Device, procedure and therapy related AEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Capel, MSc, Study Director — Sequana Medical; Christina Fotopoulou, Ph.D, Principal Investigator — Hammersmith Hospitals NHS Trust
Locations (3):
- Universitätsklinikum Leipzig, Leipzig, Germany
- Inselspital, Bern, Switzerland
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fotopoulou C, Berg T, Hausen A, Hennig R, Jalan R, Malago M, Capel J, De Gottardi A, Stirnimann G. Continuous low flow ascites drainage through the urinary bladder via the Alfapump system in palliative patients with malignant ascites. BMC Palliat Care. 2019 Dec 5;18(1):109. doi: 10.1186/s12904-019-0497-3. PMID 31805921